CLINICAL TRIAL: NCT04468633
Title: The Baerveldt Versus ClearPath Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00105781
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Baerveldt 350 implant; Ahmed ClearPath implant
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Baerveldt 350 implant (Active Comparator)
  Interventions: Device: Baerveldt 350 implant
- Ahmed ClearPath 350 implant (Active Comparator)
  Interventions: Device: Ahmed ClearPath 350 implant

INTERVENTIONS:
Device: Baerveldt 350 implant — The Baerveldt implant is an FDA-approved silicone, non-valved implant.
  Arms: Baerveldt 350 implant
Device: Ahmed ClearPath 350 implant — The Ahmed ClearPath is a non-valved glaucoma drainage device.
  Arms: Ahmed ClearPath 350 implant

SUMMARY:
This is a randomized prospective study of post-operative surgical outcomes and complication rates in patients with a Baerveldt 350 implant vs the Ahmed ClearPath implant. Each subject will be randomized to the Baerveldt group or ClearPath group at the time of consent for the study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with age at screening ≥ 18 years and ≤ 90 years
* Inadequately controlled glaucoma
* Valve-less aqueous shunt as the planned surgical procedure
* Patients with primary glaucomas or pseudoexfoliation, pigmentary and traumatic glaucoma with a previous failed trabeculectomy or other intraocular surgery included.
* Primary tubes included
* Investigators to recruit consecutively all eligible patients from their clinics.
* Superotemporal or inferonasal placement of the tube
* Capable and willing to provide consent

Exclusion Criteria:

* NLP
* Unable/unwilling to provide informed consent
* Unavailable for regular follow up
* Previous cyclodestructive procedure
* Prior scleral buckling procedure or other external impediment to supratemporal drainage device implantation
* Presence of silicone oil
* Vitreous in the anterior chamber sufficient to require a vitrectomy
* Uveitic glaucoma
* Neovascular glaucoma
* Nanophthalmos
* Sturge-Weber syndrome or other conditions associated with elevated episcleral venous pressure
* Procedure combined with other surgery
* Any abnormality other than glaucoma in the study eye that could affect tonometry.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Herndon, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Duke Eye Center (Durham, NC, USA) and its satellite locations from December 2020 to June 2023.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Started | 37; 37 eyes | 39; 39 eyes
Completed | 33; 33 eyes | 39; 39 eyes
Not Completed | 4; 4 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (9.9) | 69.6 (11.8) | 70.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 15 | 24 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 13 | 11 | 24
  Race: Black | 24 | 27 | 51
  Race: Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Time Frame: Baseline, Day 1, Week 1, Week 4, Week 6, Month 3, Month 6, and Year 1
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 33 | 39
Number analyzed (eyes) | 33 | 39
mmHg
  Baseline | 21.7 (7.1) | 22.4 (6.7)
  Day 1: number analyzed (Participants) | 32 | 38
  Day 1: number analyzed (eyes) | 32 | 38
  Day 1 | 14.9 (12.1) | 12.6 (10.5)
  Week 1: number analyzed (Participants) | 32 | 37
  Week 1: number analyzed (eyes) | 32 | 37
  Week 1 | 10.7 (5.8) | 11.5 (6.5)
  Week 4: number analyzed (Participants) | 32 | 36
  Week 4: number analyzed (eyes) | 32 | 36
  Week 4 | 16.0 (8.1) | 15.6 (9.2)
  Week 6: number analyzed (Participants) | 32 | 35
  Week 6: number analyzed (eyes) | 32 | 35
  Week 6 | 16.2 (9.7) | 12.1 (5.4)
  Month 3: number analyzed (Participants) | 32 | 33
  Month 3: number analyzed (eyes) | 32 | 33
  Month 3 | 16.5 (6.6) | 12.8 (6.5)
  Month 6: number analyzed (Participants) | 32 | 31
  Month 6: number analyzed (eyes) | 32 | 31
  Month 6 | 14.0 (4.3) | 12.5 (4.5)
  Month 12: number analyzed (Participants) | 31 | 30
  Month 12: number analyzed (eyes) | 31 | 30
  Month 12 | 14.1 (4.3) | 11.4 (3.9)
Statistical Analysis 1: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Baseline; Test type: Other; p = 0.687, t-test, 2 sided
Statistical Analysis 2: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Day 1; Test type: Other; p = 0.384, t-test, 2 sided
Statistical Analysis 3: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Week 1; Test type: Other; p = 0.597, t-test, 2 sided
Statistical Analysis 4: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Week 4; Test type: Other; p = 0.860, t-test, 2 sided
Statistical Analysis 5: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Week 6; Test type: Other; p = 0.032, t-test, 2 sided
Statistical Analysis 6: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Month 3; Test type: Other; p = 0.026, t-test, 2 sided
Statistical Analysis 7: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Month 6; Test type: Other; p = 0.172, t-test, 2 sided
Statistical Analysis 8: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Year 1; Test type: Other; p = 0.010, t-test, 2 sided

2. Primary Outcome: Number of Participants Who Experienced a Complication
Time Frame: Up to Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 37 | 39
Participants | 13 | 4

3. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Time Frame: Baseline, Day 1, Week 1, Week 4, Week 6, Month 3, Month 6, and Year 1
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 33 | 39
Number analyzed (eyes) | 33 | 39
LogMAR
  Baseline | 0.40 (0.53) | 0.56 (0.71)
  Day 1: number analyzed (Participants) | 32 | 38
  Day 1: number analyzed (eyes) | 32 | 38
  Day 1 | 0.71 (0.66) | 1.09 (0.86)
  Week 1: number analyzed (Participants) | 32 | 36
  Week 1: number analyzed (eyes) | 32 | 36
  Week 1 | 0.65 (0.68) | 1.03 (0.87)
  Week 4: number analyzed (Participants) | 32 | 36
  Week 4: number analyzed (eyes) | 32 | 36
  Week 4 | 0.45 (0.50) | 0.71 (0.84)
  Week 6: number analyzed (Participants) | 32 | 35
  Week 6: number analyzed (eyes) | 32 | 35
  Week 6 | 0.49 (0.68) | 0.71 (0.86)
  Month 3: number analyzed (Participants) | 31 | 33
  Month 3: number analyzed (eyes) | 31 | 33
  Month 3 | 0.44 (0.68) | 0.77 (0.88)
  Month 6: number analyzed (Participants) | 32 | 31
  Month 6: number analyzed (eyes) | 32 | 31
  Month 6 | 0.46 (0.68) | 0.71 (0.80)
  Year 1: number analyzed (Participants) | 31 | 30
  Year 1: number analyzed (eyes) | 31 | 30
  Year 1 | 0.36 (0.55) | 0.72 (0.76)

4. Secondary Outcome: Number of Individual Eyedrop Medications That the Patient is on (Prescribed and Actually Taking)
Time Frame: Baseline, Day 1, Week 1, Week 4, Week 6, Month 3, Month 6, and Year 1
Population: Participants with data collected at each timepoint.
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 33 | 39
medications
  Baseline | 2.7 (1.1) | 2.7 (1.5)
  Day 1: number analyzed (Participants) | 32 | 38
  Day 1 | 0.6 (0.8) | 0.7 (1.2)
  Week 1: number analyzed (Participants) | 32 | 37
  Week 1 | 0.8 (1.2) | 0.9 (1.4)
  Week 4: number analyzed (Participants) | 32 | 36
  Week 4 | 1.1 (1.3) | 1.2 (1.5)
  Week 6: number analyzed (Participants) | 32 | 35
  Week 6 | 1.4 (1.3) | 1.1 (1.3)
  Month 3: number analyzed (Participants) | 32 | 33
  Month 3 | 1.5 (1.2) | 1.4 (1.3)
  Month 6: number analyzed (Participants) | 32 | 31
  Month 6 | 2.0 (1.3) | 1.7 (1.4)
  Month 12: number analyzed (Participants) | 31 | 30
  Month 12 | 2.3 (1.2) | 1.6 (1.5)

5. Secondary Outcome: Change in Humphrey Visual Field (HVF)
Description: The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. A positive value indicates an increase in visual field while a negative value indicates a decrease.
Time Frame: Baseline and Year 1
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 27 | 25
dB | 2.81 (9.58) | 4.72 (13.55)
Statistical Analysis 1: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Test type: Other; p = 0.759, Wilcoxon rank sum test

6. Secondary Outcome: Change in Thickness of the Cornea as Measured by Pachymetry
Description: Pachymetry is an ophthalmological test that measures the thickness of the cornea.
Time Frame: Baseline and Year 1
Population: Participants with data collected at both timepoints.
Measure: Median (Standard Deviation); unit: µm
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 28 | 26
µm | 12.18 (25.86) | 25.96 (57.79)
Statistical Analysis 1: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Test type: Other; p = 0.603, Wilcoxon rank sum test

7. Other Pre Specified Outcome: Quality of Life, as Measured by Glaucoma Related Quality of Life 15 Questionnaire
Time Frame: Year 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quality of Life, as Measured by Glaucoma Symptom Scale
Time Frame: Year 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Quality of Life, as Measured by Glaucoma Utility Index
Time Frame: Year 1
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Self-report Dysesthesia Scale Questionnaire
Time Frame: Baseline and Year 1
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Motility Exam (Hess Screen Test)
Description: If patient is binocular
Time Frame: Baseline and Year 1
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Motility Exam (Worth 4-dot)
Description: If patient is binocular
Time Frame: Baseline and Year 1
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Motility Exam (Stereo Test)
Description: If patient is binocular
Time Frame: Baseline and Year 1
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Motility Exam (9 Gaze Photos)
Time Frame: Baseline and Year 1
Reporting Status: Not Posted

15. Secondary Outcome: Change in Retinal Nerve Fiber Layer (RNFL)
Description: The retinal nerve fiber layer (RNFL) is formed by retinal ganglion cell axons, which collect the visual impulses that begin with the rods and cones.
Time Frame: Baseline and Year 1
Population: Participants with data collected at both timepoints.
Measure: Median (Standard Deviation); unit: µm
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
Number analyzed (Participants) | 27 | 25
µm | 2.81 (9.58) | 4.72 (13.55)
Statistical Analysis 1: Comparison: Baerveldt 350 Implant vs Ahmed ClearPath 350 Implant; Test type: Other; p = 0.833, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Baerveldt 350 Implant | Ahmed ClearPath 350 Implant
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/39
Other Adverse Events (participants affected / at risk) | 9/37 | 8/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baerveldt 350 Implant (N=37) | Ahmed ClearPath 350 Implant (N=39)
Myocardial infarction (heart attack) (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baerveldt 350 Implant (N=37) | Ahmed ClearPath 350 Implant (N=39)
Surgical failure (Surgical and medical procedures) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT04468633/Prot_SAP_000.pdf